CLINICAL TRIAL: NCT03358186
Title: A Multi-center Study on Investigating the Surgical Treatment Effect of Periprosthetic Femur Fracture After Hip Arthroplasty
Brief Title: Investigation on the Surgical Treatment Effect of Periprosthetic Femur Fracture After Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, pengzhang, Department of orthopaedics and trauma, Peking University People's Hospital
Other Study IDs: csg-pffh
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Periprosthetic Fractures
Keywords: Periprosthetic Fractures; Arthroplasty; Surgical procedures
MeSH Terms: conditions — Periprosthetic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- revision of periprosthetic fracture: patients with surgically treated periprosthetic femur fracture
  Interventions: Procedure: surgically treated periprosthetic femur fracture

INTERVENTIONS:
Procedure: surgically treated periprosthetic femur fracture — patients with surgically treated periprosthetic femur fracture

SUMMARY:
To Investigate the Surgical Treatment effect of Periprosthetic Femur Fracture After Hip Arthroplasty

DETAILED DESCRIPTION:
In the study，155 patients from multiple center with periprosthetic femur fracture after hip arthroplasty are planned to be recruited. All the patients are treated surgically according to Vancouver classification，and their fracture union，pain in fracture site and lower extremity length are evaluated at 6 months and 1 year postoperatively．Also Harris scores are used to assess hip function at the 2 time points.

ELIGIBILITY:
Inclusion Criteria:

patients with periprosthetic femur fracture after hip arthroplasty

Exclusion Criteria:

Severe complications after surgery

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with surgically treated periprosthetic femur fracture after hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
fracture union | 1 year after surgery
  fracture union from X-ray

SECONDARY OUTCOMES:
hip function | 1 year after surgery
  Harris Hip Score
pain in fracture site | 1 year after surgery
  VAS score
lower extremity length | 1 year after surgery
  The lengths of injured lower extremity

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No